CLINICAL TRIAL: NCT07084545
Title: EPIC: Evaluation of the Postoperative Cataract Surgery Outcomes in Patients With Prior Corneal Laser Vision Correction Implanted With the CT LUCIA Intraocular Lens Protocol GPAS-SAS-023-4
Brief Title: Evaluation of Cataract Surgery Outcomes in Patients With Prior Laser Vision Correction Implanted With the CT LUCIA Lens
Status: Recruiting | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: GPAS-SAS-023-4
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Visual Outcomes Following Cataract Surgery in Patients With Prior Myopic Corneal Laser Vision Correction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CT LUCIA 621P IOL Implantation Group: Subjects with prior myopic corneal laser vision correction undergoing bilateral cataract surgery implanted with the CT LUCIA 621P intraocular lens. All subjects will be followed prospectively to assess postoperative visual and refractive outcomes.
  Interventions: Device: CT LUCIA 621P Intraocular Lens Implantation

INTERVENTIONS:
Device: CT LUCIA 621P Intraocular Lens Implantation — The intervention consists of bilateral implantation of the CT LUCIA 621P intraocular lens (IOL) during routine cataract surgery in patients with a history of myopic corneal laser vision correction. The CT LUCIA 621P IOL is an approved, single-piece, hydrophobic acrylic lens designed to provide improved visual quality and refractive stability. Implantation is performed following each investigator's standard surgical procedures, including preoperative preparation, operative technique, and postoperative care. IOL power calculation uses the ZEISS Cataract Workflow platform with the VERACITY system and Barrett True-K with TK formula, incorporating the VERION Optical Coherence (VOC) technology.

SUMMARY:
This is a prospective, Phase IV, post-approval observational study evaluating postoperative outcomes in patients with a history of myopic corneal laser vision correction (LVC) undergoing bilateral cataract surgery with implantation of the CT LUCIA 621P intraocular lens (IOL). Up to 30 subjects (60 eyes) will be enrolled across up to three U.S. investigational sites. The study will assess visual and refractive outcomes, including biometry, manifest refraction, and patient-reported visual function over a 3-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age or older.
2. Previous cornea LVC surgery performed at least 1 year before the implantation of the CT LUCIA 621P IOL, such as Laser-Assisted Intrastromal Keratomileusis (LASIK), Laser-Assisted Subepithelial Keratectomy (LASEK), Photorefractive Keratectomy (PRK) or Small Incision Lenticule Extraction (SMILE) for mild to moderate myopia, with or without astigmatism (up to, but not including, -6.0 D sphere in any meridian for myopic ablations.
3. Presenting for planned bilateral cataract extraction with in-the-bag posterior chamber IOL implantation, via phacoemulsification with or without femtosecond laser assisted cataract surgery (FLACS). Astigmatism management techniques, such as Astigmatic Keratotomy (AK), may be utilized during cataract surgery to target a predicted postoperative cylinder less than 0.75 D.
4. Clear intraocular media other than cataract (i.e., no hyphema, vitreous hemorrhage).
5. No visual acuity limiting corneal or retinal pathologies.
6. Able to and having provided written informed consent and a signed Health Insurance Portability and Accountability Act (HIPAA) form.
7. Availability, willingness, ability, and sufficient cognitive awareness to comply with study examination procedures and the schedule for study visits and evaluations.

Exclusion Criteria:

1. Implantation of an IOL other than the CT LUCIA 621P in one or both eyes.
2. Eyes with preoperative anterior corneal astigmatism of ΔTK ≥1.00 D as measured by the IOLMaster 700 or with greater than 0.75 D predicted post-operative astigmatism at the spectacle plane.
3. Visual field loss which has an impact on visual acuity.
4. Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that would confound visual acuity measurement.
5. Subjects with surgical complications in whom a CT LUCIA 621P IOL cannot be implanted in either eye.
6. Eyes with irregular corneal astigmatism, epithelial basement membrane dystrophy, chronic dry eye requiring continual treatment, underwent more than one LVC procedure in one or both eyes, or complications from the previous LVC which required additional surgical intervention.
7. Subjects with planned ocular surgery during the study (except Nd:YAG capsulotomy is permitted).
8. History of acute or chronic disease, pathology, illness, or ocular trauma that would, in the opinion of the investigator, confound results.
9. Current diagnosis of macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, amblyopia, or other chronic ocular conditions that would confound the study results.
10. A current diagnosis of moderate or severe glaucoma.
11. Patients with strabismus, forme fruste keratoconus, keratoconus or other corneal pathologies that would confound visual acuity measurement.
12. Previous radial keratotomy (RK).
13. Previous corneal keratoplasty (e.g., corneal transplant, Descemet's stripping automated endothelial keratoplasty (DSAEK), lamellar keratoplasty).
14. Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy).
15. Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate under mesopic/scotopic conditions).
16. Capsular or zonular abnormalities or other conditions that may affect the postoperative centration or tilt of the lens (e.g., pseudoexfoliation syndrome).
17. Usage of contact lenses during study participation.
18. Concurrent participation in another device investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective Phase IV post-approval study will enroll up to 30 subjects (60 eyes) at up to three U.S. sites. Eligible adults undergoing bilateral cataract surgery with the CT LUCIA 621P IOL will be enrolled after providing informed consent. Subjects must meet all protocol-defined inclusion and exclusion criteria. Those with complete baseline and Month 3 postoperative biometry and manifest refraction data in both eyes will be considered evaluable. All implanted eyes will be included in safety and efficacy analyses.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mean Prediction Error (PE) | 3 months postoperatively
  The average difference between postoperative manifest refraction spherical equivalent (MRSE) and predicted MRSE based on IOLMaster 700 with Barrett True-K with TK formula.
Median Prediction Error (PE) | 3 months postoperatively
  The median difference between postoperative MRSE and predicted MRSE based on IOLMaster 700 with Barrett True-K with TK formula.
Absolute Prediction Error (PE) | 3 months postoperatively
  The absolute value of the difference between postoperative MRSE and predicted MRSE based on IOLMaster 700 with Barrett True-K with TK formula.
Percentage of Eyes Within ±0.25 D of Predicted MRSE | 3 months postoperatively
  The proportion of eyes achieving postoperative MRSE within ±0.25 D of the predicted MRSE based on IOLMaster 700 with Barrett True-K with TK formula.
Percentage of Eyes Within ±0.50 D of Predicted MRSE | 3 months postoperatively
  The proportion of eyes achieving postoperative MRSE within ±0.50 D of the predicted MRSE based on IOLMaster 700 with Barrett True-K with TK formula.
Percentage of Eyes Within ±1.00 D of Predicted MRSE | 3 months postoperatively
  The proportion of eyes achieving postoperative MRSE within ±1.00 D of the predicted MRSE based on IOLMaster 700 with Barrett True-K with TK formula.

SECONDARY OUTCOMES:
Corrected Distance Visual Acuity (CDVA) | 3 months postoperatively
  Monocular and binocular postoperative corrected distance visual acuity measured by standard methods.
Uncorrected Distance Visual Acuity (UDVA) | 3 months postoperatively
  Monocular and binocular postoperative uncorrected distance visual acuity.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Berkeley Eye Center, Sugar Land, Texas
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No